CLINICAL TRIAL: NCT03505957
Title: A Feasibility Study Evaluating the Use of SafeBreak Vascular in the Geriatric Trauma Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lineus Medical (Industry)
Collaborators: Washington University School of Medicine (Other); Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: v001 03.09.2018
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: IV Dislodgement
Keywords: IV Dislodgement

STUDY DESIGN:
Intervention Model Description: SafeBreak Vascular works with all IVs. The study participants will have SafeBreak Vasculars installed in all of their existing IV lines or new IV lines that are installed during their enrollment in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SafeBreak Vascular Intervention (Experimental): Every study participant will have SafeBreak Vasculars installed in each of their IV lines.
  Interventions: Device: SafeBreak Vascular

INTERVENTIONS:
Device: SafeBreak Vascular — SafeBreak Vascular will be installed in all the IV lines of consenting participants for up to 7 days.
  Other Names: SafeBreak

SUMMARY:
SafeBreak Vascular is a medical device indicated for fluid flow control during the administration of IV fluids/medication to the patient's vascular system and to aid in the prevention of unintended disruption and dislodgment of IVs. SafeBreak Vascular may be used for any hospitalized patient with gravity tubing or IV pumps, for intermittent infusion or continuous infusion.The primary objective of this study is to determine if the delivery of IV medications and/or fluids with SafeBreak Vascular functions with the same reliability as current standard IV tubing.

DETAILED DESCRIPTION:
Study participants will have a SafeBreak Vascular installed in each of their existing or newly installed IV lines. The clinical literature shows in prospective observational studies that a mean of 9.2% of patients dislodge their peripheral IVs. SafeBreak Vascular is a medical device designed to aid in the prevention of unintended disruption and dislodgement of IVs, such as peripheral IVs, peripherally inserted central lines, central lines, etc. SafeBreak IV will be installed in each IV line between the study participant's catheter and the IV tubing that goes to the IV bag or IV pump. When a harmful force is placed on the IV line, SafeBreak Vascular is designed to separate so that the harmful force is removed from the line and IV dislodgement is prevented. SafeBreak Vascular has a valve in each end of the device. Upon separation, each valves closes, stopping the flow of fluid. The primary objective of the study is to determine if the delivery of IV medications and/or fluids with SafeBreak Vascular functions with the same reliability as current standard IV tubing. The number of IV dislodgements and IV restarts will be recorded. The study will also collect data for analysis concerning the following:

* device design characteristics
* certain human factors (patient or operator) associated with the use of the device
* the impact of this device usage on clinician workflow
* any unknown safety concerns
* obtain preliminary data for use in designing a subsequent pivotal study of the device.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric trauma patients (> or equal to age 55)
* Participants able to provide informed consent or have a legally authorized representative (LAR) provide consent
* The patients must have IV access (existing central venous catheter, peripherally inserted central catheter, or peripheral IV's) or need IV access
* The patients must be at least 55 years of age.

Exclusion Criteria:

* Unable to obtain informed consent or without an available LAR to provide surrogate informed consent
* Age less than or equal to 54
* Patient on comfort care only
* Predicted to have less than 24 hours survival
* Patient enrolled in an investigational drug or device study at the time of enrollment
* Investigator discretion that patient is not suitable for the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
IV dislodgement rate | Up to 7 days
  Compare the study intervention's rate of IV dislodgement to the clinical literature's prospective observational studies that have a mean dislodgement of 17.5% and median of 9.2%.

SECONDARY OUTCOMES:
IV restarts | Up to 7 days.
  Comparison of the study's intervention to the clinical literature's rates for IV failure, which is 46% of IVs fail before the end of their intended use
Device related adverse events | Up to 7 days
  Collection of any adverse events related to SafeBreak Vascular

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bochicchio, RN, MS, Study Director — Washington University School of Medicine; Stacey Reese, RN, MS, Study Director — Washington University of St. Louis
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kornbau C, Lee KC, Hughes GD, Firstenberg MS. Central line complications. Int J Crit Illn Inj Sci. 2015 Jul-Sep;5(3):170-8. doi: 10.4103/2229-5151.164940. PMID 26557487
- [Background] Helm RE, Klausner JD, Klemperer JD, Flint LM, Huang E. Accepted but unacceptable: peripheral IV catheter failure. J Infus Nurs. 2015 May-Jun;38(3):189-203. doi: 10.1097/NAN.0000000000000100. PMID 25871866